CLINICAL TRIAL: NCT06053099
Title: A Prospective Cohort Study to Evaluate Molecular pRognostic Factors and Resistance Mechanisms to Osimertinib in Adjuvant Treatment of Completely Resected pIB-IIIA Non-small Cell Lung Carcinoma With Common EGFR Mutations (L858R and Del19)
Acronym: ROSIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IFCT-2202
Record Dates: First submitted 2023-08-18; First posted 2023-09-25 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Non Small Cell Lung Cancer; EGFR Activating Mutation; EGFR DEL19; EGFR L858R
Keywords: IFCT; NSCLC; Adjuvant Osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plasma ctDNA and FFPE blocks (Experimental)
  Interventions: Other: Plasma ctDNA; Other: FFPE blocks

INTERVENTIONS:
Other: Plasma ctDNA — * Plasma ctDNA before surgery (optional)
  * Plasma ctDNA post-surgery : 4 to 8 weeks post-surgery, before starting adjuvant chemotherapy (if given) and before starting adjuvant osimertinib (if given)
  * Plasma ctDNA every 6 months
  * Plasma ctDNA at relapse
Other: FFPE blocks — * Surgery FFPE blocks
  * FFPE blocks at relapse (optional)

SUMMARY:
IFCT-2202 ROSIE study aims to incorporate a broad-panel centralized NGS testing at baseline in all patients with completely resected NSCLC with common EGFR mutation after confirmation of an optimal preoperative extension assessment and with a centralized review of the quality of the surgical excision. Furthermore, the IFCT-2202 ROSIE study also aims to study the molecular events associated with relapse on, or after osimertinib exposure, that should result in the opportunity to accede to optimal treatment in case of metastatic relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent.
2. Age ≥ 18 years.
3. Pre-surgical disease evaluation including brain MRI/CT-scan and total body PET-FDG CT-scan prior to surgery.
4. Histologically complete anatomical resection (R0) of stage pIB-IIIA (pTNM 8th edition) NSCLC.
5. Presence of a common EGFR mutation (Del19 or L858R).
6. Archival tumour tissue FFPE blocks from surgery available for centrally molecular analyses.
7. Patient eligible to receive osimertinib adjuvant therapy in a 3-year intent to treat decision; patients could receive if necessary adjuvant chemotherapy before starting osimertinib treatment.
8. Patient who is capable, according to the investigator, of complying with the study's requirements and restrictions.
9. Patient followed in the institution on a regular basis (every 3 to 6 months) according to standard recommendations.
10. Estimated life expectancy > 3 years.
11. Woman patients who are of childbearing potential are eligible:

    * They must have a negative pregnancy test before the first dose of osimertinib.
    * They must agree to use effective methods of contraception throughout the course of treatment and should be maintained for 2 months after the end of treatment.
12. Male subjects who are sexually active with a woman of childbearing potential are eligible if an efficacious contraception method should be used during the treatment and during the 4 months following the last dose.

Exclusion Criteria:

1. History of cancer, except for the following situations:

   Patients with history of cancer for more than 3 years are eligible if they have been treated and considered cured. Patients with history of in situ carcinoma of the cervix or non-melanoma skin carcinoma are eligible.
2. Neoadjuvant anti-cancer treatment (osimertinib and/or chemotherapy or other anti-cancer treatment).
3. Incompletely resected NSCLC (R1 or R2).
4. Any medical condition that would, according to the investigator's judgment, prevent the patient's participation in the clinical study.
5. Active infection (e.g. patients receiving treatment for infection) including hepatitis C virus (HCV) and human immunodeficiency virus (HIV), or active uncontrolled hepatitis B infection except for the situations described in APPENDIX I. Screening for chronic conditions is not required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility study | 18 months
  Number of patients included receiving osimertinib after 18 months of enrollment

SECONDARY OUTCOMES:
Incidence, nature, and severity of osimertinib-related adverse events (safety) | About 3 years
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0).

CONTACTS AND LOCATIONS:
Locations (36):
- France (36):
  - Angers - CHU, Angers
  - Bayonne - CH, Bayonne
  - Boulogne - Ambroise Paré, Boulogne
  - Lyon - URCOT, Bron
  - Caen - CHU, Caen
  - Clermont-Ferrand - CHU, Clermont-Ferrand
  - Colmar - CH, Colmar
  - Créteil - CHI, Créteil
  - Dijon - CHU Bocage, Dijon
  - Grenoble - CHU, Grenoble
  - La Roche-Sur-Yon - CH, La Roche-sur-Yon
  - Le Mans - CHG, Le Mans
  - Lille - CHU, Lille
  - Lyon - CRLCC, Lyon
  - Marseille - APHM, Marseille
  - Metz - Hôpital Robert Schuman, Metz
  - Montpellier - CHU, Montpellier
  - Montpellier - ICM, Montpellier
  - Nice - CHU, Nice
  - Orléans - CHR, Orléans
  - Paris - Bichat, Paris
  - Paris - HEGP, Paris
  - Paris - Hôpital Cochin, Paris
  - Paris - Pitié-Salpêtrière, Paris
  - Paris - Tenon, Paris
  - Pau - CHG, Pau
  - Bordeaux - CHU, Pessac
  - Poitiers - CHU, Poitiers
  - Annecy - CH, Pringy
  - Rennes - CHU, Rennes
  - Rouen - CHU, Rouen
  - Strasbourg - NHC, Strasbourg
  - Suresnes - Foch, Suresnes
  - Toulon - CHI, Toulon
  - Toulouse - CHU, Toulouse
  - Tours - CHU, Tours

IPD SHARING:
Plan to Share IPD: Undecided